CLINICAL TRIAL: NCT00562211
Title: A Single-blind, Randomized, Controlled Trial to Assess the Efficacy of a New Topical Anesthetic in Reducing Pain Associated With Venipuncture in Children.
Brief Title: Efficacy of a New Topical Anesthetic
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, i_shavit, Pediatric Emergency Department director, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2465CTIL; 2465
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2007-11

CONDITIONS: Pain
Keywords: children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: LidoDyn
- 2 (Active Comparator)
  Interventions: Drug: EMLA creme

INTERVENTIONS:
Drug: LidoDyn — Application of 2 gram of LidoDyn to the skin surface the patient's antecubital fossa 60 min prior to venipuncture
  Arms: 1
Drug: EMLA creme — Application of 2 gram of EMLA creme to the skin surface the patient's antecubital fossa 60 min prior to venipuncture
  Arms: 2

SUMMARY:
A new topical anesthetic which contains 5% lidocaine and a disinfection ingredient has been developed and is tested in this study (LidoDyn).

The study examines the efficacy of LidoDyn by comparing it with an already proven anesthetic agent (EMLA crème).

ELIGIBILITY:
Inclusion Criteria:

* Previously healthy children of whom venipuncture is needed to be performed.

Exclusion Criteria:

* History of allergic reaction to any local anesthetic.
* History of chronic disease
* Patient's condition requires urgent treatment (e.g. severe dehydration, shock)
* Active local skin infection or skin pathologic condition at the antecubital fossa
* Tattoo, surgical scar or skin condition that might interfere with skin sight assessment.
* Patient undergone venipuncture at the antecubital fossa within the pror two weeks.
* Uncooperative or exceptionally anxious patient.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Self report assessment of pain (using the Visual Analog Scale) | 60 Min+ 5-10 Min

SECONDARY OUTCOMES:
Medical staff observational assessment of pain (in a scale of 0 to 10) | 60 Min + 5-10 Min

CONTACTS AND LOCATIONS:
Overall Officials: Itai Shavit, M.D., Principal Investigator — Rambam Health Care Campus; Hadas Knaani-Levinz, M.D., Principal Investigator — Rambam Health Care Campus; Amir Hadash, M.D., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Emergency Department of the Meyer Children Hospital, Rambam Health Care Campus, Haifa, Israel